CLINICAL TRIAL: NCT04526483
Title: Safety and Efficacy of a Novel Intelligent Navigation 4K UHD 3D Endoscopic Imaging System in Laparoscopic Gastrectomy
Brief Title: L-Gastrectomy With the Intelligent Navigation 4K UHD 3D Endoscopic Imaging System
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Minimally Invasive Surgery Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LG-4K, 3D & ICG
Record Dates: First submitted 2020-08-19; First posted 2020-08-25 (Actual); Last update posted 2020-08-25 (Actual); Status verified 2020-08

CONDITIONS: Stomach Neoplasms
Keywords: Laparoscopy; Gastrectomy; 4K; 3D; lymphadenectomy
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Intervention Model Description: This is a prospective, one-arm, single-center, single-set target value clinical trial to investigate the clinical value of the Intelligent Navigation 4K UHD 3D Endoscopic Imaging System on laparoscopic gastric surgery. The trial will recruit a total of 67 participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- laparoscopic gastrectomy with Intelligent Navigation 4K UHD 3D (Experimental)
  Interventions: Device: Laparoscopic gastrectomy with Intelligent Navigation 4K UHD 3D Endoscopic Imaging System

INTERVENTIONS:
Device: Laparoscopic gastrectomy with Intelligent Navigation 4K UHD 3D Endoscopic Imaging System — Laparoscopic gastrectomy with Intelligent Navigation 4K UHD 3D Endoscopic Imaging System

SUMMARY:
This study aims to evaluate the safety, efficacy, and feasibility of the Intelligent Navigation 4K UHD 3D Endoscopic Imaging System in patients with gastric cancer.

DETAILED DESCRIPTION:
Background: Lymphadenectomy in laparoscopic gastrectomy can significantly improve the long-term survival and accuracy of the tumor staging of patients with gastric cancer. The retrieval of more lymph nodes has gradually become a trend among surgeons. However, lymphadenectomy is currently performed without the aid of visual instruments which might lead to an unknown pathological outcome and influence the prognosis of gastric cancer patients. And none of the indocyanine green (ICG) fluorescent imaging systems applied in clinical practice now is equipped with ultra-high definition (4K) or three-dimensional (3D) lens. To explore the advent of minimally invasive surgery with a conveniently switchable high-quality imaging system, we designed a new laparoscopic navigating technique that combined all the three characteristics.

Aims: This study aims to evaluate the safety, efficacy, and feasibility of the Intelligent Navigation 4K UHD 3D Endoscopic Imaging System in patients with gastric cancer.

Methods/design This is a prospective, one-arm, single-center, single-set target value clinical trial to investigate the clinical value of the Intelligent Navigation 4K UHD 3D Endoscopic Imaging System on laparoscopic gastric surgery. The trial will recruit a total of 67 participants.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with gastric cancer require surgery;
2. Without a history of abdominal surgery;
3. BMI ≤ 30 kg/m2;
4. Preoperative ECOG score is 0~1 and ASA score is I~III;
5. Having signed the Medical Informed Consent.

Exclusion Criteria:

1. Patients with metastasis or invasion of surrounding tissues;
2. Undergoing emergency operation (perforation, hemorrhage, obstruction);
3. Patients with serious medical co-morbidity (heart, lung, liver and kidney diseases) and could not tolerate laparoscopic surgery;
4. With poor incorrigible physical condition before surgery;
5. The patient who underwent gastrojejunostomy or jejunostomy;
6. The patient who refuses to accept standardized postoperative systemic therapy according to the guidelines.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Estimated)
Dates: Start 2020-10-01 (Estimated); Primary Completion 2022-10-01 (Estimated); Study Completion 2022-10-01 (Estimated)

PRIMARY OUTCOMES:
The success rate of laparoscopic gastric surgery | 24 months
  Rate of successfully performed laparoscopic gastrectomy

SECONDARY OUTCOMES:
Lymph node dissection rate | 24 months
  The numbers of lymph node dissected in the surgery

IPD SHARING:
Plan to Share IPD: Undecided